CLINICAL TRIAL: NCT05341908
Title: Prevalence of Pathogens in Synovial Fluid Obtained From Emergency Department Patients and Clinical and Laboratory Features of Patients Diagnosed With Septic Arthritis
Brief Title: Prevalence of Pathogens in Synovial Fluid Obtained From Emergency Department Patients
Status: Completed | Type: Observational
Sponsor: Olive View-UCLA Education & Research Institute (Other)
Collaborators: Biofire, Inc (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, David A. Talan, Professor of Medicine, Olive View-UCLA Education & Research Institute
Other Study IDs: 1577712
Record Dates: First submitted 2021-11-10; First posted 2022-04-22 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Septic Arthritis; Joint Infection
MeSH Terms: conditions — Arthritis, Infectious

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Synovial fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, observational study of patients presenting to the emergency departments at 9 EMERGEncy ID NET sites. The objectives of the proposed study are to:

1. Describe the range and proportion of infectious agents in synovial fluid as detected by standard C&S and investigational PCR testing, i.e., Biofire® Film Array® Bone and Joint Infection (BJI) Panel,
2. Describe the epidemiology of patients receiving diagnostic arthrocentesis and those diagnosed with septic arthritis in the emergency department (ED),
3. Determine the prevalence of septic arthritis in US ED patients presenting with an atraumatic painful swollen joint, and
4. Determine the clinical (history and physical examination) and laboratory characteristics of septic arthritis.

Study coordinators screen the ED log for adult patients presenting with joint pain and whose treating physician ordered an arthrocentesis. After confirming eligibility, study coordinators approach the patient to explain the study, and present the written consent form. If the patient agrees to participate and consent, the study coordinator completes an enrollment data collection using patient and treating physician interview to gather responses. After enrollment, the study coordinator will ensure that approximately 0.3-1.0 mL of leftover synovial fluid is saved and stored in a freezer for shipment to a central laboratory (Truman Medical Center hospital laboratory, Kansas City, MO) for testing. Approximately 30 days after enrollment, study coordinators complete an electronic medical record (EMR) review.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older;
2. diagnostic arthrocentesis in the emergency department (ED) or during hospitalization if admitted from the ED;
3. arthrocentesis and joint culture ordered; and
4. provide written consent in English or Spanish

Exclusion Criteria:

1. Unable to consent or no legal authorized representative is available; or
2. prisoner or parolee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, multicenter, observational study being conducted at 9 EMERGEncy ID NET sites, Olive View-UCLA Medical Center, Los Angeles, CA; Temple University Hospital, Philadelphia, PA; University of Mississippi Medical Center, Jackson, MS; Valleywise Medical Center, Phoenix, AZ; Truman Medical Center/U. Missouri Kansas City, Kansas City, MO; Hennepin Medical Center, Minneapolis, MN, University of New Mexico Health Sciences Center, Albuquerque, NM; University of Iowa Hospital, Iowa City, IA; and Johns Hopkins Medical Institute, Baltimore, MD. These hospitals service a mostly urban and underserved population.
  Patients presenting to the above hospital emergency departments will be approached by study team members who meet the above eligibility criteria. The target enrollment for the study is 500 participants.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of pathogens | Two years
  We will describe the prevalence of pathogens identified using PCR testing
Prevalence of septic arthritis | Two years
  We will describe the prevalence of septic arthritis among patients who have joint taps in emergency departments

SECONDARY OUTCOMES:
Clinical characteristics of septic arthritis | Two years
  We will compare clinical characteristics, such as duration of symptoms, medical history, immunocompromising conditions, vitals, and demographics between those who have septic arthritis vs. those who do not to determine if there are possible predictors
Laboratory characteristics of septic arthritis | Two years
  We will compare laboratory characteristics, such as white blood cell count, presence of crystals, gram stain, and culture results between those who have septic arthritis vs. those who do not to determine if there are possible predictors

CONTACTS AND LOCATIONS:
Locations (1):
- Olive View-UCLA Medical Center, Sylmar, California, United States

IPD SHARING:
Plan to Share IPD: No